CLINICAL TRIAL: NCT03126149
Title: A Phase 1, Randomized, Double-blind (Sponsor-open), Placebo-controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Single Escalating Oral Doses Of Pf-06667272 Under Fed And Fasted Conditions, In Healthy Adult Subjects
Brief Title: First in Human Study for PF-06667272
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C0231002; 2017-000590-36 (EudraCT Number)
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (16):
- Cohort 1_Period 1_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 1_Period 1_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Cohort 1_Period 2_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 1_Period 2_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Cohort 1_Period 3_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 1_Period 3_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Cohrot 1_Period 4_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 1_Period 4_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Cohort 2_Period 1_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 2_Period 1_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Cohort 2_Period 2_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 2_Period 2_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Cohort 2_Period 3_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 2_Period 3_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Cohort 2_Period 4_Active (Experimental): Single ascending dose of PF-06667272
  Interventions: Drug: PF-06667272
- Cohort 2_Period 4_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06667272 — Single ascending dose of PF-06667272
  Arms: Cohort 1_Period 1_Active; Cohort 1_Period 2_Active; Cohort 1_Period 3_Active; Cohort 2_Period 1_Active; Cohort 2_Period 2_Active; Cohort 2_Period 3_Active; Cohort 2_Period 4_Active; Cohrot 1_Period 4_Active
Other: Placebo — Single dose of placebo
  Arms: Cohort 1_Period 1_Placebo; Cohort 1_Period 2_Placebo; Cohort 1_Period 3_Placebo; Cohort 1_Period 4_Placebo; Cohort 2_Period 1_Placebo; Cohort 2_Period 2_Placebo; Cohort 2_Period 3_Placebo; Cohort 2_Period 4_Placebo

SUMMARY:
The current study is the first clinical trial proposed with PF-06667272. It is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of single ascending doses of PF-06667272 under fed and fasted conditions, in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential;
* Body Mass Index 17.5-30.5 kg/m2;
* Body weight >50 kg;

Exclusion Criteria:

* Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Treatment Emergent Treatment-Related Adverse Events (AEs) or other safety concerns | Baseline (Day 1, hour 0) up to 28 days after last dose of study medication
  Assessment by adverse event monitoring, 12 lead ECGs, telemetry, vital signs and clinical safety laboratory measurements.
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06667272 and PF-06818073 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for PF-06667272 and PF-06818073 (as permitted) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Maximum Observed Plasma Concentration (Cmax) for PF-06667272 and PF-06818073 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Concentration for PF-06667272 and PF-06818073 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) for PF-06667272 and PF-06818073 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Apparent Total Body Clearance (CL/F) for PF-06667272 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after apparent total body clearance is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) for PF-06667272 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0231002&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind+%28sponsor-open%29%2C+Placebo-controlled+Study+To+Assess+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Single+Escalating+Oral+Doses+Of+Pf-06667272+Under+Fed+And+Fasted+Conditions%2C+In+Healthy+Adult+Subjects